CLINICAL TRIAL: NCT07166120
Title: Precision Treatment to Promote Smoking Cessation and Survival in Oncology Patients
Acronym: PROMISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202403025; LC230570 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Smoking Cessation; Smoking; Physician's Role
Keywords: Genetics; Primary Care Physicians; Tobacco Treatment
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Intervention Model Description: Randomization occurs at the clinician level. For pragmatic concerns, the investigators expect to recruit from multiple clinics and cluster randomization of clinicians will be stratified by clinics to minimize the clinic effect. Given the stratified randomization by clinic and the possibility of an unequal number of physicians across the 2 arms (i.e., we may not have exactly 8 in each arm), the investigators aim to recruit 8 clinicians per arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Active Comparator): The arm will represent usual care in the oncology care clinics. Clinicians will receive a report designed to recommend guideline-based tobacco treatment. Patients will receive a report on guideline-based advice about smoking cessation and a brief discussion with a behavior interventionist.
  Interventions: Behavioral: Usual care
- PrecisionTx-Onc (oncology) (Experimental): Clinicians will receive PrecisionTx-Onc, an intervention designed to recommend precision tobacco treatment, adapted for oncology. Patients will receive PrecisionTx-Onc, an intervention designed to recommend precision tobacco treatment, and a brief discussion with a behavior interventionist, adapted for oncology.
  Interventions: Behavioral: Precision treatment

INTERVENTIONS:
Behavioral: Usual care — Usual care will be informed by practice guidelines (standard of care, brief advice, and guideline awareness).
  Arms: Usual Care
Behavioral: Precision treatment — Precision treatment will be informed by practice guidelines (standard of care, brief advice, and guideline awareness), plus patient-specific risk feedback and personalized tobacco treatment recommendations using patients' clinical, genetic, and biomarker information, adapted for oncology.
  Arms: PrecisionTx-Onc (oncology)

SUMMARY:
This study evaluates the feasibility and preliminary effects of precision tobacco treatment, compared to usual care, on promoting tobacco treatment in oncology patients and providers in the oncology care setting. The precision treatment intervention includes personalized tobacco treatment recommendations using the patient's clinical, genetic, and biomarker information. This intervention may increase patient receipt of tobacco treatment, patient medication use, and patient smoking abstinence at 6 months.

DETAILED DESCRIPTION:
This study aims to promote the provision and use of evidence-based tobacco treatment and patient survival by integrating precision tobacco treatment into oncology care as a novel multilevel intervention. This study builds on growing evidence that 1) precision treatment may optimize treatment effectiveness by precisely matching patients with the safest, most effective medications available and 2) precision intervention may boost the implementation and effectiveness of tobacco treatment. The multilevel precision treatment intervention to be tested-PrecisionTx-- provides the opportunity to present personalized risk, benefit, and treatment recommendation to increase clinician ordering, patient uptake, and overall effectiveness of tobacco treatment.

This study aims to understand the feasibility and preliminary effects of precision treatment over usual care and associated mechanistic and implementation outcomes. Therefore, the investigators propose a 2-arm cluster randomized controlled trial of 16 clinicians and 96 patients (~6 per clinician) from oncology care settings. Clinicians and patients will be randomized with 1:1 allocation to usual care (UC) vs. precision treatment (PT) to evaluate the effect of precision treatment on patient receipt of tobacco treatment and smoking abstinence.

In Aim 1, the investigators will develop a contextually grounded multilevel PT intervention, PrecisionTx-Onc, for oncology/hematology clinics by engaging both patients and providers. In Aim 2, the investigators will conduct a 2-arm RCT to pilot the multilevel PT intervention for feasibility and determine preliminary estimates of clinical outcomes. Preliminary data will address hypotheses that the PT vs. the UC condition will produce superior physician prescribing as measured by patient receipt of prescription, patient medication use, and patient bioverified smoking abstinence at 6 months. Additional outcomes include patient quality of life and survival.

In Aim 3, the investigators will explore mechanisms of behavior change and implementation outcomes. The investigators will explore 1) mechanisms (e.g., outcome expectancies, perceived risk/benefit, and withdrawal suppression) underlying the effect of PT, and 2) implementation outcomes to evaluate its potential for scaling, using the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework.

Primary outcomes include patient receipt of tobacco treatment, patient use of tobacco treatment, and patient smoking abstinence. Secondary outcomes include patient receipt of recommended medication, patient medication adherence, patient quality of life, patient survival, and additional patient smoking cessation outcomes. Mechanistic outcomes include clinician level (perceived benefit, outcome expectancy), clinician-patient interaction (self-efficacy), patient-level (perceived risk, outcome expectancy, withdrawal suppression, adverse events). Implementation outcomes will be evaluated based on the RE-AIM framework.

The study is an innovative paradigm shift from a traditional treatment model to precision treatment that includes both metabolic and genetic markers to motivate and guide tobacco treatment for both clinicians and patients, integrated within oncology care. This study will test the impact of a multilevel precision treatment intervention on improving tobacco treatment and health outcomes in oncology care.

ELIGIBILITY:
Eligibility Criteria for Clinicians:

* Clinician from participating oncology/hematology clinic
* At least 18 years of age
* Can speak and understand English

Inclusion Criteria for Patients:

* Patient at participating clinic
* Age 18-89 years
* Current smoking (average cigarettes per day ≥5)
* Can speak and understand English
* Willing to consider medication to help reduce craving or smoking such as nicotine patch, lozenge, or varenicline

Exclusion Criteria for Patients:

* Active use of smoking cessation medication (within the past 30 days)
* Receipt of smoking cessation medication or prescription for smoking cessation medication (within the past 30 days)
* Having a contradiction for cNRT or varenicline (allergic reactions, current cardiac problems, pregnancy)
* Patients who were deemed by the investigator to be ineligible for participation in the trial

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient receipt of tobacco treatment medication for smoking cessation | 6 months post-intervention
  This will be quantified by the proportion of enrolled patients who receive cessation medication.
Patient use of cessation medication | 6 months post-intervention
  This will be quantified by the proportion of patients taking any cessation medication from time of enrollment through 6 months post-intervention.
Patient smoking abstinence | 6 months post-intervention
  This will be quantified by the proportion of patients who smoke with bioverified point-prevalent abstinence at 6 months.

SECONDARY OUTCOMES:
Patient quality of life | 6 and 12 months post-intervention
  Quality of life measure will be measured using European Organization for Research and Treatment of Cancer Quality of life Questionnaire-Core 30 (EORTC QLQ-C30). All of the scales and single-item range in score from 0-100. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents high quality of life, but a high score for a symptom scale / item represents a high level of symptomatology/problems.
Patient survival | 6 and 12 months post-intervention
  Probability of survival from the start of intervention
Patient receipt of recommended tobacco treatment | 6 months post-intervention
  This will be quantified by the proportion of enrolled patients who received recommended cessation medication.
Patient medication adherence | 6 months post-intervention
  This will be quantified by the proportion of medication taken among medication prescribed.
Patient smoking abstinence among treated | 6 months post-intervention
  This will be quantified by the proportion of smokers with bioverified point-prevalence abstinence among those receiving cessation medication.
Abstinence Outcomes Across Multiple Time Points | From intervention through 12 months post-intervention
  The outcome measures abstinence (self-reported no smoking (not even a puff of a cigarette) for at least 7 days prior to the assessment) over these time points.
Smoking quantity across multiple time points | From intervention through 12 months post-intervention
  The outcome measures smoking quantity (self-reported average cigarettes smoked per day for the past 30 days prior to the assessment) over these time points.
Quit attempts | 6 and 12 months post-intervention
  This outcome measures the number of quit attempts in the past 30 days prior to the assessment over these time points.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Shiun Chen, ScD, M.D., MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu